CLINICAL TRIAL: NCT02608645
Title: Evaluation of Perceptions, Knowledge and Compliance With tHE Guidelines for Secondary Prevention in Real Life Practice: A Survey on the Under-treatment of hypercholeSterolemia (EPHESUS Trial)
Brief Title: A Survey on the Under-treatment of hypercholeSterolemia (EPHESUS Trial)
Acronym: EPHESUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Murat Biteker, Assoc. Prof. Mugla Sitki Kocman University, Muğla Sıtkı Koçman University
Other Study IDs: EPHESUS trial
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, within the secondary prevention group patients ( diabetes mellitus, coronary artery disease, peripheral artery disease, who have had events atherosclerotic cerebrovascular ) , statin use requirement , patients compliance and reaching target LDL-cholesterol levels (according to European guidelines ) will be evaluated.

DETAILED DESCRIPTION:
In the majority of patients treated with lipid lowering agents are not under control in accordance with the lipids manual. In this study, within the secondary prevention group patients ( diabetes mellitus, coronary artery disease, peripheral artery disease, who have had events atherosclerotic cerebrovascular ) , statin use requirement , patients compliance and reaching target LDL-cholesterol levels (according to European guidelines ) will be evaluated.

The investigators' aim is to determine the role of education and knowledge in reaching target LDL cholesterol levels in these patients. İn addition , the investigators want to emphasize in high-risk patients who are receiving or not receiving cholesterol-lowering treatment what is their target values , (LDL < 100 mg / dL and high -risk patients with LDL < 70 mg / dL in very high-risk patients ) and to determine what is the rate of patients and to the importance of reaching their target cholesterol levels. İn addition ,to evaluate the patients habits of the using statin dose .After screening , physician treatment decisions and reasons will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease (acute coronary syndromes, post- myocardial infarction patients, who have a history of percutaneous coronary intervention , history of coronary artery by-pass graft )
* Patients with carotid artery lesions or peripheral artery disease ,
* Type 2 diabetes mellitus patients

Exclusion Criteria:

* acute coronary syndrome in last 1 month
* pregnancy or the first 6 months postpartum
* ICU patients or emergency patients...etc.(other than polyclinic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving lipid-lowering therapy within the secondary prevention group in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The number of patients with secondary prevention group receiving appropriate lipid lowering therapy | 2 months

REFERENCES:
- [Derived] Dogan V, Basaran O, Ozlek B, Celik O, Ozlek E, Cil C, Ozdemir IH, Rencuzogullari I, Ozpamuk Karadeniz F, Bekar L, Aktas M, Resulzade MM, Kalcik M, Aksan G, Cinier G, Halli Akay K, Mert KU, Biteker M, Kayikcioglu M. Evaluation of perceptions, knowledge and compliance with guidelines in real-life practice: A survey on the under-treatment of hypercholesterolemia. Turk Kardiyol Dern Ars. 2019 Oct;47(7):599-608. doi: 10.5543/tkda.2019.39293. PMID 31582673
- [Derived] Dogan V, Basaran O, Ozlek B, Celik O, Ozlek E, Mert KU, Rencuzogullari I, Mert GO, Dogan MM, Biteker M, Kayikcioglu M. Rationale, design, and methodology of the Evaluation of Perceptions, Knowledge, and Compliance with the Guidelines in Real Life Practice: A Survey on the Under-treatment of Hypercholesterolemia. Turk Kardiyol Dern Ars. 2018 Jan;46(1):47-53. doi: 10.5543/tkda.2017.73861. PMID 29339691